CLINICAL TRIAL: NCT00593073
Title: Use of Novel Tailored Reminders in Rural Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Kimberly K. Engelman, PhD, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 10174; 1R21CA121907-01 (NIH)
Record Dates: First submitted 2007-12-31; First posted 2008-01-14 (Estimated); Last update posted 2008-09-12 (Estimated); Status verified 2008-09

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Tailored Reminder Message
  Interventions: Behavioral: Electronic tailored messaging
- 2 (Experimental): General Reminder Message
  Interventions: Behavioral: General Reminder Message

INTERVENTIONS:
Behavioral: Electronic tailored messaging — Tailored CRC message based on patient screening barriers, preferences and attitudes and reminder to get screened.
  Arms: 1
Behavioral: General Reminder Message — General CRC health education message and reminder to get screened.
  Arms: 2

SUMMARY:
Effective programs are needed that can overcome barriers to CRC screening among persons in rural communities. There is good evidence to suggest that a program employing patient activation and tailoring to address the specific concerns of individuals will be an effective model for addressing CRC screening underutilization for rural residents. In this study, we propose to test such a model among rural primary care patients, a group that has, to date, received little attention. We will also bolster how tailored messaging is traditionally conducted by using a tailored informational flyer format that uses physicians as the message source to increase message saliency. This study will help to assess how a relatively low-cost, disseminable technology can effectively circumvent the "systems problems" endemic in rural primary care. This project will lay the groundwork in practice based research network clinics for future intervention studies which operationalize office and community-based technology to help rural primary care patients make informed health decisions and engage in healthy lifestyle behaviors.

DETAILED DESCRIPTION:
Screening for colorectal cancer (CRC) remains severely underutilized. Although simple reminders are modestly effective in enhancing preventive care utilization, they are not widely utilized. Even if used widely, the effectiveness of simple reminders is limited, leaving nearly half of patients without screening. One explanation for this is that simple reminders do not address the barriers and resources of the patients and physicians they are designed to prompt. In this study, we will examine the impact on CRC screening of a reminder system that uses the physician as the message source and is tailored to the physician screening preferences and patient-reported characteristics, CRC screening-related barriers, status and CRC susceptibility. This intervention will be compared to a standard CRC health education and screening reminder system.

Touch screen 'Healthy Living' computer kiosks will be placed in 16 Kansas Physicians Engaged in Prevention Research (KPEPR) Network primary care practices. The kiosk program will screen for eligible participants who are at least 50 years of age and not up-to-date with CRC screening and guide eligible participants through a computerized Colorectal Cancer Assessment (CRCA). Kiosk participants will be randomized into either a general CRC health education + screening reminder message (GRM) (N=640) or a patient and physician-tailored CRC + screening reminder message (TRM) (N=640). Immediately upon completion of the CRCA, GRM participants will receive a brief informational flyer with general CRC health education messages and a reminder to get screened routinely for CRC. Participants in the TRM arm will receive an informational flyer that contains messages that are tailored to patient CRC screening barriers, preferences, and attitudes and physician screening preferences (guided by CRC screening options that are available within the local community) in addition to a reminder to get screened for CRC. A 90-day telephone follow-up will assess participant compliance with CRC screening recommendations, participant discussion with their physician regarding CRC screening, and patient satisfaction.

This study will use a novel patient- and physician- tailored messaging approach to promote colorectal cancer screening utilization. This study will help to assess how a practice-based computerized patient activation approach can effectively circumvent the "systems problems" endemic in rural primary care and lay the groundwork for future computer-based primary care intervention studies to help patients make informed health decisions and engage in healthy lifestyle behaviors.

ELIGIBILITY:
Inclusion Criteria:

* 50 years of age or older
* at average risk for colorectal cancer
* not up to date with colorectal cancer screening

Exclusion Criteria:

* Younger than 50 years of age
* at high risk for colorectal cancer
* up to date with colorectal cancer screening

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 707 (Actual)
Dates: Start 2005-07; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Baseline assessment while waiting to see primary care physician and 90-day follow-up telephone survey. | Baseline, 90 Days

SECONDARY OUTCOMES:
Follow-up survey to assess participant discussion of colorectal cancer with their healthcare provider and compliance with CRC screening | 90 Days

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly K. Engelman, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States